CLINICAL TRIAL: NCT07276438
Title: MRI- or CT-Guidance and Online Adaptation With Stereotactic Radiotherapy for Prostate Cancer (MANTICORE)
Brief Title: Image-Guidance and Online Adaptation With Stereotactic Body Radiation Therapy for the Treatment of Localized Prostate Cancer, MANTICORE Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Viewray Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-000781; NCI-2025-07701 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-000781 (Other: UCLA / Jonsson Comprehensive Cancer Center); P30CA016042 (NIH); R37CA292795 (NIH)
Record Dates: First submitted 2025-12-01; First posted 2025-12-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Localized Prostate Adenocarcinoma; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Investigator
Masking Description: This block size will be blinded to the radiation oncology research team when enrolling a patient. The arm allocation will be masked until after the screening/baseline data are entered and filled out in Research Electronic Data Capture (REDCap) (no anticipation of the group assignment will be possible).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm 1 (non-adaptive SBRT) (Active Comparator): Patients undergo MRI or CT-guided SBRT without daily plan adaptation once every other day or QD for a total of 5 treatments over 18 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo MRI and CT during screening and blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Radiation: CT-guided Stereotactic Body Radiation Therapy; Procedure: Magnetic Resonance Imaging; Radiation: MRI-guided Stereotactic Body Radiation Therapy; Other: Survey Administration
- Arm 2 (adaptive SBRT) (Experimental): Patients undergo MRI or CT-guided SBRT with daily plan adaptation once every other day or QD for a total of 5 treatments over 18 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo MRI and CT during screening and blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Radiation: CT-guided Stereotactic Body Radiation Therapy; Other: Inter-fraction Adaptation of Treatment Plan; Procedure: Magnetic Resonance Imaging; Radiation: MRI-guided Stereotactic Body Radiation Therapy; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Radiation: CT-guided Stereotactic Body Radiation Therapy — Undergo CT-guided SBRT
  Other Names: Computed Tomography-Guided Stereotactic Body Radiation Therapy; CT-guided SBRT
Other: Inter-fraction Adaptation of Treatment Plan — Undergo daily plan adaptation
  Other Names: Inter-fraction adaptation
  Arms: Arm 2 (adaptive SBRT)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Radiation: MRI-guided Stereotactic Body Radiation Therapy — Undergo MRI-guided SBRT
  Other Names: Magnetic Resonance Imaging-guided Stereotactic Body Radiation Therapy; MR-guided SBRT; MRI-guided SBRT
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial studies the side effects of image-guidance and online adaptation with stereotactic body radiation therapy (SBRT) for the treatment of patients with prostate adenocarcinoma that has not spread to other parts of the body (localized). Image-guided SBRT is a standard treatment for localized prostate cancer. This treatment uses imaging of the cancer within the body to define and localize the area to be treated with the radiation. Imaging can be obtained using either computed tomography (CT), magnetic resonance imaging (MRI), or a combination of the two. Typically, with SBRT, a radiation plan is developed based on the CT or MRI images obtained before treatment begins and adjustments are not made to the plan during treatment. However, anatomy can be different from day-to-day which may cause radiation to be delivered to the normal surrounding structures and possibly more side effects. During image-guided SBRT with online adaptation, the initial radiation plan is designed similarly; however, when the patient presents for radiation, the attending radiation oncologist, a dosimetrist, and a medical physicist "re-optimize" the radiation plan using the current anatomy of the day, meaning the changes in bladder and prostate size/shape are taken into account. The initial plan and the re-optimized plan are then compared, and the plan that has the optimal balance between delivering a tumor killing dose of radiation and minimizing radiation dose to normal surrounding structures is delivered. Image-guidance and online adaptation with SBRT may lower side effects and be a safer way to treat localized prostate adenocarcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether daily, real-time adaptive SBRT to the prostate improves acute patient-reported genitourinary (GU) toxicity when compared with conventional, non-adaptive SBRT to the prostate for localized prostate cancer.

SECONDARY OBJECTIVES:

I. To determine whether there are differences in the acute, patient-reported other toxicity following daily, real-time adaptive versus conventional, non-adaptive SBRT for localized prostate cancer.

II. To determine whether there are chronic differences in patient-reported quality of life (QOL) outcomes following daily, real-time adaptive versus conventional, non-adaptive SBRT for localized prostate cancer.

III. To determine whether there are differences in the acute and late physician-scored GU and gastrointestinal (GI) toxicity following daily, real-time adaptive versus conventional, non-adaptive SBRT for localized prostate cancer.

IV. To determine whether there are differences in the 5-year biochemical recurrence-free survival (BCRFS) following daily, real-time adaptive versus conventional, non-adaptive SBRT for localized prostate cancer.

CORRELATIVE OBJECTIVE:

I. To correlate patient-reported and physician-scored toxicity with a commercially available genetic biomarker (PROSTOX trademark, MiraDx, Los Angeles, CA).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients undergo MRI or CT-guided SBRT without daily plan adaptation once every other day or once daily (QD) for a total of 5 treatments over 18 days in the absence of disease progression or unacceptable toxicity.

ARM 2: Patients undergo MRI or CT-guided SBRT with daily plan adaptation once every other day or QD for a total of 5 treatments over 18 days in the absence of disease progression or unacceptable toxicity.

Additionally, all patients undergo MRI and CT during screening and blood sample collection throughout the trial.

After completion of study treatment, patients are followed up at months 1, 3, 6, 9, 12, 24, 36, 48, and 60.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Histologically confirmed, clinically localized adenocarcinoma of the prostate
* Staging workup as recommended by the National Comprehensive Cancer Network (NCCN) on the basis of risk grouping

  * Advanced imaging studies (i.e. prostate-specific membrane antigen [PSMA] positron emission tomography [PET]/CT and fluciclovine PET/CT scan) can supplant a bone scan if performed first
* No evidence of metastatic disease in lymph nodes above the bifurcation of the renal arteries, or in bones or visceral organs (nodal disease identified on a PSMA PET/CT scan below the bifurcation of the renal arteries are amenable)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* No indication for urgent or emergent radiation
* Written informed consent obtained from participant or participant's legal representative and ability for participant to comply with the requirements of the study

Exclusion Criteria:

* Patients with neuroendocrine or small cell carcinoma of the prostate
* Patients with any evidence of distant metastases except that evidence of lymphadenopathy below the level of the renal arteries can be deemed locoregional per the discretion of the investigator
* Prior cryosurgery, high-intensity focused ultrasound (HIFU), brachytherapy, or other ablative treatments of the whole prostate
* Prior pelvic radiotherapy
* History of Crohn's disease, ulcerative colitis, or ataxia telangiectasia
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the participant or the quality of the data

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute clinically relevant decline in the urinary irritative/obstructive subdomain of the Expanded Prostate Cancer Index Composite Short Form Questionnaire (EPIC-26) | From start of stereotactic body radiation therapy (SBRT) to 90 days following SBRT
  A clinically relevant decrement in the EPIC-26 urinary irritative/obstructive domain is defined as greater than 14 points. Will compare the proportion of patients with a clinically relevant in genitourinary EPIC-26 urinary irritative/obstructive subdomain within 90 days of study therapy via a simple binomial test for differences in proportions. A more granular analysis will be based on the cumulative incidence method will be used to summarize risk of clinically relevant decline and Fine-Gray test will be used to compare cumulative incidences between the two arms. The analysis population includes all randomized subjects based on intent-to-treat principle. Point estimates as well as the associated 95% confidence intervals will be reported. Will also be evaluated using a multivariable analysis adjusted for variables including a simultaneous integrated boost, use of nodal radiotherapy, and use of hydrogel spacers.

SECONDARY OUTCOMES:
Acute change in EPIC-26 scores | From start of SBRT to 90 days following SBRT
  Will be represented by changes from baseline in the urinary incontinence, bowel, sexual function, and hormone/vitality domains. Changes will be analyzed with respect to whether they represent clinically relevant differences, defined as greater than 18, 12, and 24 points for urinary incontinence, bowel, and sexual domains, respectively. Analysis will be performed using a restricted maximum likelihood (REML)-based mixed models repeated measures (MMRM) approach. The model will include the fixed categorical effects of treatment, time, and treatment-by-time interaction, as well as the other fixed baseline covariates. An unstructured covariance structure will be used to model the within-patient errors. The Kenward-Roger approximation will be used to estimate denominator degrees of freedom. The analysis of acute changes in the bowel domain of the EPIC-26 instrument will be stratified for use of hydrogel spacers or not.
Acute change in International Prostate Symptom Score (IPSS) | From start of SBRT to 90 days following SBRT
  The numerical change from baseline, as well as the raw score at any given timepoint, will be extracted and reported descriptively; an absolute change of ≥ 15 points on IPSS will be considered a clinically relevant change. Analysis will be performed using a REML-based MMRM approach. The model will include the fixed categorical effects of treatment, time, and treatment-by-time interaction, as well as the other fixed baseline covariates. An unstructured covariance structure will be used to model the within-patient errors. The Kenward-Roger approximation will be used to estimate denominator degrees of freedom.
Acute change in Sexual Health Inventory for Men (SHIM) scores | From start of SBRT to 90 days following SBRT
  The numerical change from baseline, as well as the raw score at any given timepoint, will be extracted and reported descriptively; an absolute change of ≥ 10 points on the SHIM will be considered a clinically relevant change. Analysis will be performed using a REML-based MMRM approach. The model will include the fixed categorical effects of treatment, time, and treatment-by-time interaction, as well as the other fixed baseline covariates. An unstructured covariance structure will be used to model the within-patient errors. The Kenward-Roger approximation will be used to estimate denominator degrees of freedom.
Chronic change in EPIC-26 scores | From start of SBRT to 60 months following SBRT
  Will be represented by changes from baseline in the urinary incontinence, bowel, sexual function, and hormone/vitality domains. Changes will be analyzed with respect to whether they represent clinically relevant differences, defined as greater than 18, 12, and 24 points for urinary incontinence, bowel, and sexual domains, respectively. Analysis will be performed using a REML-based MMRM approach. The model will include the fixed categorical effects of treatment, time, and treatment-by-time interaction, as well as the other fixed baseline covariates. An unstructured covariance structure will be used to model the within-patient errors. The Kenward-Roger approximation will be used to estimate denominator degrees of freedom. The analysis of chronic changes in the bowel domain of the EPIC-26 instrument will be stratified for use of hydrogel spacers or not.
Chronic change in IPSS | From start of SBRT to 60 months following SBRT
  The numerical change from baseline, as well as the raw score at any given timepoint, will be extracted and reported descriptively; an absolute change of ≥ 15 points on IPSS will be considered a clinically relevant change. Analysis will be performed using a REML-based MMRM approach. The model will include the fixed categorical effects of treatment, time, and treatment-by-time interaction, as well as the other fixed baseline covariates. An unstructured covariance structure will be used to model the within-patient errors. The Kenward-Roger approximation will be used to estimate denominator degrees of freedom.
Chronic change in SHIM scores | From start of SBRT to 60 months following SBRT
  The numerical change from baseline, as well as the raw score at any given timepoint, will be extracted and reported descriptively; an absolute change of ≥ 10 points on the SHIM will be considered a clinically relevant change. Analysis will be performed using a REML-based MMRM approach. The model will include the fixed categorical effects of treatment, time, and treatment-by-time interaction, as well as the other fixed baseline covariates. An unstructured covariance structure will be used to model the within-patient errors. The Kenward-Roger approximation will be used to estimate denominator degrees of freedom.
Incidence of physician-scored acute grade ≥ 2 genitourinary (GU) and gastrointestinal (GI) toxicities | From start of SBRT to 90 days following SBRT
  As assessed using Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 scale. The analysis of both acute and late GI toxicity will be stratified for use of hydrogel spacers or not and by use of nodal radiotherapy or not, if event rate permits this analysis.
Incidence of physician-score late grade ≥ 2 GU and GI toxicities | From start of SBRT to 60 months following SBRT
  As assessed using CTCAE v 5.0 scale. The analysis of both acute and late GI toxicity will be stratified for use of hydrogel spacers or not and by use of nodal radiotherapy or not, if event rate permits this analysis.
Biochemical recurrence-free survival | Up to 60 months
  Will be estimated by the Kaplan-Meier method as well as descriptively (mean, standard deviation, median, first and third quartiles, minimum, maximum), with biochemical recurrence defined as serum prostate-specific antigen (PSA) levels that are 2 ng/mL higher than the nadir PSA achieved after SBRT. Figures showing the Kaplan-Meier estimates will also be presented. Death of any cause will be treated as a competing risk.

CONTACTS AND LOCATIONS:
Overall Officials: Amar W. Kishan, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States